CLINICAL TRIAL: NCT06577792
Title: Lobectomy-First Versus Lymphadenectomy-First Surgical Approach on Long-Term Survival in Operable Non-Small Cell Lung Cancer Patients: A Prospective, Multi-Center, Randomized Study
Brief Title: Lobectomy-First vs. Lymphadenectomy-First for Operable NSCLC (LOFTY)
Acronym: LOFTY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Tianjin Medical University Cancer Institute and Hospital (Other); RenJi Hospital (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); First Affiliated Hospital of Jinan University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Shanghai Changzheng Hospital (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Suining Central Hospital (Other); The Affiliated Hospital of Xuzhou Medical University (Other); The General Hospital of Eastern Theater Command (Other); Fujian Medical University Union Hospital (Other); First Affiliated Hospital of Kunming Medical University (Other); Fujian Provincial Hospital (Other); Tianjin Chest Hospital (Other); Sichuan Cancer Hospital and Research Institute (Other); Tang-Du Hospital (Other); Shandong Provincial Hospital (Other Government); Gansu Provincial Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Wuhan TongJi Hospital (Other); The Affiliated Hospital of Qingdao University (Other); West China Hospital (Other); Jiangsu Cancer Institute & Hospital (Other); Dongguan People's Hospital (Other Government); First People's Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Hao-Xian Yang, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SL-B2022-443; ChiCTR2300068586 (Registry Identifier: Chinese Clinical Trial Registry)
Record Dates: First submitted 2024-07-08; First posted 2024-08-29 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non-small cell lung cancer; Lobectomy; Lymphadenectomy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lobectomy-First group (Other): Patients with operable NSCLC received lobectomy first then received lymphadenectomy for surgical treatment.
  Interventions: Procedure: Lobectomy-First
- Lymphadenectomy-First group (Other): Patients with operable NSCLC received lymphadenectomy first then received lobectomy for surgical treatment.
  Interventions: Procedure: Lymphadenectomy-First

INTERVENTIONS:
Procedure: Lobectomy-First — During the surgical treatment for patients with NSCLC, thoracic surgeons should perform lobectomy first, and then perform lymphadenectomy next.
  Arms: Lobectomy-First group
Procedure: Lymphadenectomy-First — During the surgical treatment for patients with NSCLC, thoracic surgeons should perform lymphadenectomy first, and then perform lobectomy next.
  Arms: Lymphadenectomy-First group

SUMMARY:
During the surgery for non-small cell lung cancer (NSCLC), lymphadenectomy or lobectomy are performed first, different surgeons have different choices. Oncology textbooks require dissecting distant lymph nodes (LNs) first and then dissecting nearby LNs. According to this requirement, thoracic surgeons should first perform lymphadenectomy and then lobectomy. Unfortunately, there is no high-level evidence to prove which surgical sequence is more beneficial to the long-term survival of NSCLC patients. In this multi-center randomized controlled trial (RCT), patients with stage I-II NSCLC were enrolled as the research object to determine which surgical sequence (lymphadenectomy-first vs. lobectomy-first) is better for the short-term and long-term outcomes in NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 80 years old;
2. The first clinical diagnosis before surgery was non-small cell lung cancer, including adenocarcinoma, squamous cell carcinoma, large cell carcinoma, and other unknown types;
3. Clinical stage T1-2N0-1 (cI-II): Maximum diameter of tumor <= 5 cm and short diameter of mediastinal lymph node <= 1cm in thin layer computed tomography (CT);
4. The patient's physical condition is able to tolerate lobectomy: (1) Goldman index 0-1; (2) Predicted forced expiratory volume in 1s (FEV1) >= 40% and diffusing capacity of the lung for carbon monoxide (DLCO) >= 40%; (3) Total bilirubin <= 1.5 upper limit of normal; (4) Alanine aminotransferase (ALT)/Aspartate aminotransferase (AST) <= 2.5 upper limit of normal; (5) Creatinine <= 1.25 upper limit of normal and creatinine clearance rate (CCr) >= 60 ml/min;
5. Performance status of Eastern Cooperative Oncology Group (ECOG) = 0-1;
6. All relevant examinations were completed within 28 days before the operation;
7. Patients who understand this study and have signed an approved Informed Consent.

Exclusion Criteria:

1. Patients who have undergone anti-tumor therapy (radiotherapy, chemotherapy, targeted therapy, immunotherapy) before surgery;
2. Patients with previous medical history of other malignant tumors or combined with second primary cancer at the time of enrollment;
3. Patients who meet all of the following criteria are eligible for sublobar resection (segment/wedge resection): (1) Ground glass opacity (GGO) with a solid component <= 50%; (2) The largest diameter of nodule is <= 2 cm; (3) The nodule is located in the outer third of the lung field;
4. Patients with preoperative diagnosis of pure GGO;
5. Patients with previous medical history of unilateral thoracotomy;
6. Women who are pregnant or breastfeeding;
7. Patients with active bacterial or fungal infection that is difficult to control;
8. Patients with serious psychosis;
9. Patients with a history of severe heart disease, heart failure, myocardial infarction or angina pectoris in the past 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
5-year disease-free survival (DFS) | 5 years after surgery
  The disease-free survival rate 5 years after surgery

SECONDARY OUTCOMES:
5-year overall survival (OS) | 5 years after surgery
  The overall survival rate 5 years after surgery
3-year disease free survival (DFS) | 3 years after surgery
  The disease-free survival rate 3 years after surgery
3-year overall survival (OS) | 3 years after surgery
  The overall survival rate 3 years after surgery
Intraoperative blood loss | During the surgery
  Total blood loss during the surgery
Conversion rate | During the surgery
  The number of cases converted to thoracotomy in a group divided by the total number of included cases in this group
Perioperative complications rate | The day of surgery, 2/4/8/12/26/52 weeks after surgery
  The number of cases in a group with perioperative complications divided by the total number of included cases in this group
Operative death rate | 30/90 days after surgery
  The number of cases in a group died within 30/90 days after surgery divided by the total number of cases in this group
Postoperative hospital stays | Between the date of surgery and the date of discharge, assessed up to 30 days
  The number of days between the date of surgery and the date of discharge
Postoperative pain score | Daily after surgery for up to 7 days and at weeks 2/4/8/12/26/52 after discharge
  The degree of pain after surgery was measured using Numerical Rating Scale (NRS). The patient is asked to make three pain ratings, corresponding to current, best and worst pain experienced over the past 24 hours on a scale of 0 (no pain) to 10 (worst pain imaginable). The average of the 3 ratings was used to represent the patient's level of pain over the previous 24 hours
R0 rate | Postoperative in-hospital stay up to 30 days
  The number of cases in a group received complete resection divided by the total number of cases in this group
Operative time | During the surgery
  The total time from skin to skin and the time of each step
Chest tube duration | Postoperative in-hospital stay up to 30 days
  The number of days between the date of surgery and the date of chest tube removal
The numbers of circulating tumor cell (CTC)/circulating tumor DNA (ctDNA) before and after operation | During the surgery
  3ml of peripheral arterial blood was drawn before surgery and immediately after chest closure, and then CTC/ctDNA was isolated by differential centrifugation for quantitative measurement
Acesodyne (Grade III) dose | Postoperative in-hospital stay up to 30 days
  The total amount of morphine used by the patient during the postoperative hospital period
Total cost of hospitalization | From the date of admission to the date of discharge, assessed up to 30 days
  The total medical cost of the patient from admission to discharge
The number of resected lymph nodes | Postoperative in-hospital stay up to 30 days
  The number of resected lymph nodes were calculated according to the official pathological report after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hao-Xian Yang, M.D., Principal Investigator — Sun Yat-sen University
Locations (26):
- China (26):
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - Dongguan People's Hospital, Dongguan, Guangdong
  - First People's Hospital of Foshan, Foshan, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Wuhan TongJi Hospital, Wuhan, Hubei
  - Wuhan Union Hospital, China, Wuhan, Hubei
  - Jiangsu Cancer Institute & Hospital, Nanjing, Jiangsu
  - The General Hospital of Eastern Theater Command, Nanjing, Jiangsu
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Tang-Du Hospital, Xi'an, Shaanxi
  - Shandong Provincial Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - RenJi Hospital, Shanghai, Shanghai Municipality
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital and Research Institute, Chengdu, Sichuan
  - West China Hospital, Chengdu, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fan HR, Yang MZ, Yan XL, Chen XB, Gou YJ, You J, Lin JB, Zhou HN, Zhang H, Chen WS, Zhang N, Tang H, Lin YB, Leng XF, Qian XZ, Yi J, Su XD, Cai SW, Gu WQ, Peng ZM, Du W, Yang H, Mei JD, Sun DQ, Liao YD, Liao HY, Qiu B, Ma GW, Jiao WJ, Wang W, Wang Y, Zhao ZR, Liu QW, Sun TY, Li M, Yang HX. Lobectomy-first versus lymphadenectomy-first on long-term survival for operable non-small cell lung cancer: protocol of LOFTY trial. Trials. 2025 Dec 29;26(1):581. doi: 10.1186/s13063-025-09285-9. PMID 41462323
- See also: This clinical trial has been registered in Chinese Clinical Trial Registry with a registration number as ChiCTR2300068586 — https://www.chictr.org.cn/bin/project/edit?pid=178449